CLINICAL TRIAL: NCT01977482
Title: A Phase IIB, Randomized, Blinded, Dose-ranging, Active-controlled, Parallel-group, Multi-center Study to Evaluate the Dose Response Relationship of GSK1278863 Over the First 4 Weeks of Treatment and Evaluate the Safety and Efficacy of GSK1278863 Over 24 Weeks in Hemodialysis-Dependent Subjects With Anemia Associated With Chronic Kidney Disease Who Switch From Recombinant Human Erythropoietin
Brief Title: Evaluation of Dose Response Relationship, Safety and Efficacy of GSK1278863 in Hemodialysis-dependent Subjects With Chronic Kidney Disease Associated Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113633
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Anaemia
Keywords: hemoglobin; recombinant human erythropoietin; Chronic kidney disease; hemodialysis; pharmacokinetics; erythropoiesis stimulating agents; Anemia; GSK1278863
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- GSK1278863 4 mg (Experimental): Subjects will take GSK1278863 4 mg blinded once daily (OD) orally for 4 weeks with a glass of water. From Week 4, study medication will continue to be administered OD and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: GSK1278863
- GSK1278863 6 mg (Experimental): Subjects will take GSK1278863 6 mg blinded OD orally for 4 weeks with a glass of water. From Week 4, study medication will continue to be administered OD and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: GSK1278863
- GSK1278863 8 mg (Experimental): Subjects will take GSK1278863 8 mg blinded OD orally for 4 weeks with a glass of water. From Week 4, study medication will continue to be administered OD and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: GSK1278863
- GSK1278863 10 mg (Experimental): Subjects will take GSK1278863 10 mg blinded OD orally for 4 weeks with a glass of water. From Week 4, study medication will continue to be administered OD and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: GSK1278863
- GSK1278863 12 mg (Experimental): Subjects will take GSK1278863 12 mg blinded OD orally for 4 weeks with a glass of water. From Week 4, study medication will continue to be administered OD and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: GSK1278863
- Control (Active Comparator): Subjects will take GSK1278863 matching placebo blinded OD orally for 4 weeks with a glass of water. From Week 4, rhEPO will be administered and the dose will be adjusted based on Hgb levels dose every 4 weeks till Week 24.
  Interventions: Drug: Placebo; Drug: rhEPO

INTERVENTIONS:
Drug: GSK1278863 — Film coated tablets containing 1 mg, 2 mg, 5 mg, or 25 mg of GSK1278863
  Arms: GSK1278863 10 mg; GSK1278863 12 mg; GSK1278863 4 mg; GSK1278863 6 mg; GSK1278863 8 mg
Drug: Placebo — Matching placebo tablet for GSK1278863
  Arms: Control
Drug: rhEPO — rhEPO will be procured from local market
  Arms: Control

SUMMARY:
This study is intended to evaluate the dose-response relationship of GSK1278863 over the first 4 weeks of treatment and evaluate the safety and efficacy of GSK1278863 over 24 weeks to maintain hemoglobin (Hgb) level in hemodialysis-dependent (HDD) subjects with anemia associated with chronic kidney disease (CKD) who are switched from a stable dose of recombinant human erythropoietin (rhEPO). The data generated will enable selection of the starting dose(s) and optimize dose adjustment regimen(s) for Phase 3 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects are eligible if they meet all of the inclusion criteria below:
* General criteria
* Age: >=18 years of age. (Week -4 verification only)
* Gender: Female and male subjects. (Week -4 verification only) Females: If of childbearing potential, must agree to use one of the approved contraception methods, from Screening until completion of the Follow-up Visit OR of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy, or oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) 23.0-116.3 International units per liter (IU/L) and estradiol <=10 picomole per liter (pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 weeks must elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method;
* Q-T Interval Corrected for Heart Rate (QTc): Bazett's Correction of QT Interval (QTcB) <470 millisecond (msec) or QTcB <480 msec in subjects with bundle branch block. There is no QTc inclusion criterion for a subject with a predominantly paced rhythm.
* CKD-related criteria
* Dialysis frequency: On hemodialysis (HD) three to five times weekly for at least 4 weeks prior to Week -4 Screening through Week 4. NOTE: Combination methods including hemofiltration (HF) or ultrafiltration (UF) with HD are allowed. However, the type of dialysis (HD, hemodiafiltration (HDF) or UF) should not change during the study.
* Dialysis adequacy: A single-pool dialyzer clearance multiplied by dialyzer time divided by volume of distribution of urea (Kt/Vurea) of >=1.2 based on a historical value obtained within the prior month in order to ensure the adequacy of dialysis. If Kt/Vurea is not available, then an average of the last 2 values of urea reduction ratio (URR) of at least 65%. NOTE: Only needs confirming at Week -4.
* Hemoglobin: Baseline Hgb of 9.0-11.5 g/dL (may rescreen in a minimum of 2 weeks).
* Stable rhEPO dose: Using the same rhEPO (epoetins or their biosimilars, or darbepoetin) with total weekly doses varying by no more than 50% during the 4 weeks prior to Week -4. At Day 1 (randomization), confirm that total weekly doses varied by no more than 50% during the screening period.
* Iron replacement therapy: Subjects may be on stable maintenance oral or IV (<=100 mg/week) iron supplementation. If subjects are on oral or IV iron, then doses must be stable for the 4 weeks prior to Week -4, during the screening phase, and through the first 4 weeks after Randomization.

Exclusion Criteria:

* Subjects are not eligible if they meet any of the exclusion criteria below:
* CKD-related criteria
* Dialysis modality: Planned change from HD to peritoneal dialysis within the study time period.
* Renal transplant: Pre-emptive or scheduled renal transplant.
* High rhEPO dose: An epoetin dose of >=360 IU/Kg/Week IV or >=250 IU/kg/week subcutaneous (SC) or darbepoetin dose of >=1.8 microgram (µg)/Kg/Week IV or SC within the prior 8 weeks through Day 1 (randomization).
* Use of methoxy polyethylene glycol epoetin beta within the prior 8 weeks through Day 1 (randomization).
* Laboratory test-based criteria (Week -4 verification only)
* Vitamin B12: At or below the lower limit of the reference range (may rescreen in a minimum of 8 weeks).
* Folate: <2.0 nanogram (ng)/mL (<4.5 nanomole (nmol)/L) (may rescreen in a minimum of 4 weeks).
* Ferritin: <100 ng/mL (<100 Micrograms per liter).
* Transferrin saturation (TSAT): Outside of the reference range.
* Cardiovascular disease-related criteria
* Myocardial infarction or acute coronary syndrome: Within the 8 weeks prior to Screening through Day 1 (randomization).
* Stroke or transient ischemic attack: Within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Heart failure: Class III/IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system diagnosed prior to Week -4 Screening through Day 1 (randomization); Symptomatic right heart failure diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Hypertension: Defined using pre-dialysis vitals (Week -4, Day 1) of diastolic blood pressure (DBP) >100 millimeters of mercury (mmHg) or systolic blood pressure (SBP) >170 mmHg.
* Thrombotic disease: History of thrombotic disease (e.g., venous thrombosis such as deep vein thrombosis or pulmonary embolism, or arterial thrombosis such as new onset or worsening limb ischemia requiring intervention), except vascular access thrombosis, within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Other disease-related criteria
* Ophthalmology disease: Meeting any ophthalmologic-related exclusion criteria determined at the Screening ophthalmology exam.
* Inflammatory disease: Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Hematological disease: Any hematological disease including those affecting platelets, white or red blood cells (e.g. sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia and thalassemia), coagulation disorders (e.g., antiphospholipid syndrome, Protein C or S deficiency), or any other cause of anemia other than renal disease diagnosed prior to Week -4 Screening through Day 1 (randomization).
* Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) > 2.0 x upper limit of normal (ULN) or total bilirubin > 1.5 x ULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participation in the study. NOTE: Those with Hepatitis B or Hepatitis C are eligible provided these exclusions are not met.
* Major surgery: Major surgery (excluding vascular access surgery) within the prior 8 weeks, during the Week -4 Screening phase or planned during the study.
* Transfusion: Blood transfusion within the prior 8 weeks, during the Week -4 Screening phase or an anticipated need for blood transfusion during the study.
* GI Bleeding: Evidence of actively bleeding peptic, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within the 8 weeks prior to Week -4 Screening through Day 1 (randomization).
* Acute infection: Clinical evidence of acute infection or history of infection requiring intravenous (IV) antibiotic therapy within the 8 weeks prior to Week -4 Screening through Day 1 (randomization). NOTE: IV antibiotics as prophylaxis are allowed.
* Malignancy: Subjects with a history of malignancy within the prior 5 years, who receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders); with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to Week -4 Screening through Day 1 (randomization).
* Concomitant medication and other Investigational Product-related criteria
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
* Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from Week -4 Screening until the Follow-up Visit.
* Prior investigational product exposure: The Subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days from Week -4 Screening through Day 1 (randomization).
* General health-related criteria
* Other Conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the Investigator considers would put the subject at unacceptable risk.
* Pregnancy or Lactation: Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test OR women who are lactating at Week -4 Screening or during the trial.
* Other Eligibility Criteria Considerations
* Laboratory eligibility criteria will be assessed according to the central laboratory results for the screening samples.
* Subjects who fail screening may be rescreened as soon as the investigator feels they may have become eligible. However, an individual subject may not rescreen more than twice. There is no predetermined amount of time that the investigator needs to wait to rescreen a previously ineligible subject, except those excluded for Hgb or folate who may only rescreen in 2 and 4 weeks, respectively, and those excluded for Vitamin B12 who may rescreen in 8 weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-11-01; Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (99):
- United States (16):
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Dimas, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Farmington, Missouri
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
- Australia (5):
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Czechia (5):
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Louny
  - GSK Investigational Site, Most
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Sokolov
- Denmark (2):
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
- France (4):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Paris
- Germany (7):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Demmin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Esztergom
  - GSK Investigational Site, Pécs
- Japan (7):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamagata
- Norway (4):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
- Poland (4):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Zabrze
- Russia (8):
  - GSK Investigational Site, Kaluga
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnogorsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Mytischi
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- South Korea (6):
  - GSK Investigational Site, Anyang-Si Gyeonggi-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (11):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
- Sweden (4):
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- United Kingdom (7):
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Dorchester
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Oxford

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were hemodialysis-dependent with anemia associated with chronic kidney disease who were switched from a stable dose of recombinant human erythropoietin (rhEPO).
Pre-assignment Details: A total of 216 participants with a stable hemoglobin (Hgb) between 9.0-11.5 grams (g)/deciliter (dL) (France sites only: 10.0-11.5 g/dL) were randomized.
Groups:
- Control: Participants received placebo once daily for the first 4 weeks and thereafter received open label rhEPO as required to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- GSK1278863 4 mg: Participants received GSK1278863 4 milligrams (mg) once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- GSK1278863 6 mg: Participants received GSK1278863 6 mg once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- GSK1278863 8 mg: Participants received GSK1278863 8 mg once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- GSK1278863 10 mg: Participants received GSK1278863 10 mg once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- GSK1278863 12 mg: Participants received GSK1278863 12 mg once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
Period: Overall Study
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Started | 39 | 39 | 40 | 39 | 40 | 19
Completed | 36 | 30 | 35 | 35 | 37 | 14
Not Completed | 3 | 9 | 5 | 4 | 3 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other-Protocol-defined Stopping Criteria | 0 | 3 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 3 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- GSK1278863 4 mg: Participants received GSK1278863 4 mg once daily for the first 4 weeks and thereafter, if necessary the dose was adjusted every four weeks to achieve Hgb within the range of 10.0-11.5 g/dL for the remaining 20 weeks.
- Total: Total of all reporting groups
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg | Total
Number analyzed (Participants) | 39 | 39 | 40 | 39 | 40 | 19 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 59.7 (18.74) | 58.7 (13.33) | 63.5 (14.00) | 60.1 (10.36) | 55.4 (15.50) | 59.9 (13.26) | 59.5 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 12 | 15 | 17 | 8 | 80
  Male | 26 | 24 | 28 | 24 | 23 | 11 | 136
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 23 | 28 | 28 | 28 | 31 | 12 | 150
  African American | 7 | 4 | 5 | 3 | 4 | 4 | 27
  Asian | 7 | 6 | 7 | 7 | 5 | 3 | 35
  Other | 2 | 1 | 0 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hgb) at Week 4
Description: Baseline Hgb value was the average of three Hgb values taken during screening period at Week (W) -4, W-2 and Day 1. Change from Baseline in Hgb was calculated as W4 value minus the Baseline value. To model the dose-response relationship a four-parameter Emax model was used. The dose response dataset was based on all non-missing data collected up to W4. Participants (par.) who had a Week 2 Hgb measurement, but a missing Week 4 Hgb measurement were included with a change from Baseline at Week 4 value imputed as twice the change from Baseline at Week 2. E0 is the expected Hgb change from Baseline for a par. receiving placebo and experiencing the average Hgb Baseline observed in the study. Emax is the expected Hgb change from Baseline for a par. receiving the highest dose above which no further increase in response can be achieved. ED50 is the dose that attains the intermediate response. Gamma is the slope parameter. Alpha is the coefficient of the model covariate for centred Baseline.
Time Frame: Baseline (Week -4, Week-2 and Day 1) and Week 4
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: grams (g)/deciliter (dL)
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 39 | 39 | 40 | 39 | 40 | 19
grams (g)/deciliter (dL) | -0.64 (0.829) | -0.24 (0.989) | 0.08 (1.131) | 0.42 (0.796) | 0.64 (1.177) | 0.61 (1.245)
Statistical Analysis 1: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; E0 (g/dL) = -0.664, 95% CI 2-sided [-0.960 to -0.387] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 2: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; ED50 (milligrams[mg]) = 33.531, 95% CI 2-sided [15.566 to 48.948] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 3: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Emax (g/dL) = 5.234, 95% CI [2.691 to 7.940] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 4: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Gamma = 1.145, 95% CI 2-sided [0.748 to 1.738] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 5: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Var = 1.012, 95% CI 2-sided [0.840 to 1.234] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 6: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Alpha = -0.206, 95% CI 2-sided [-0.397 to -0.014] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 7: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Minimally Effective Dose (MED) (mg) = 0.418, 95% CI 2-sided [0.000 to 2.342] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 8: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Dose that achieves a change of -0.25g/dL = 2.423, 95% CI 2-sided [0.000 to 4.150] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 9: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Target Dose (TD) (mg) = 4.406, 95% CI 2-sided [2.544 to 5.995] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 10: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Dose that achieves a change of 0.25 g/dL = 6.430, 95% CI 2-sided [4.698 to 8.010] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 11: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Dose that achieves a change of 0.5 g/dL = 8.542, 95% CI 2-sided [6.931 to 10.523] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 12: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Dose that achieves a change of 0.75 g/dL = 10.800, 95% CI 2-sided [9.024 to 14.004] — Posterior median and 95% credibility intervals were estimated using Bayesian methods
Statistical Analysis 13: Comparison: Control vs GSK1278863 4 mg vs GSK1278863 6 mg vs GSK1278863 8 mg vs GSK1278863 10 mg vs GSK1278863 12 mg; Test type: Superiority or Other; Dose that achieves a change of 1 g/dL = 13.248, 95% CI 2-sided [10.891 to 18.916] — Posterior median and 95% credibility intervals were estimated using Bayesian methods

2. Secondary Outcome: Hgb Concentration at Week 24
Description: Hgb values measured at Week 24 are presented.
Time Frame: Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 24 | 18 | 27 | 26 | 24 | 11
g/dL | 10.56 (0.974) | 10.29 (0.864) | 10.54 (1.010) | 10.63 (1.099) | 10.28 (0.856) | 10.70 (0.867)

3. Secondary Outcome: Percentage of Time Within, Below, and Above Hgb Target Range Between Weeks 20 and 24
Description: The percentage of time in Hgb target range between Weeks 20 and 24 for a participant was calculated by dividing the total number of days that Hgb was within the target range (10.0 to 11.5 g/dL) while on treatment during Weeks 20 to 24 (using linear interpolation) by the total number of days the participant remained on treatment during the defined period. Similarly, percentage of time above Hgb target range and percentage of time below Hgb target range were calculated.
Time Frame: Week 20 to Week 24
Population: ITT population. Only participants with data available at specific timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 31 | 22 | 28 | 27 | 25 | 14
Percentage of days
  Percentage of time within target range | 54.59 (42.044) | 74.77 (38.797) | 57.38 (40.505) | 37.46 (41.775) | 48.97 (42.490) | 55.23 (40.350)
  Percentage of time above target range | 24.65 (38.556) | 6.89 (22.137) | 17.18 (30.446) | 33.15 (42.856) | 18.27 (33.698) | 26.88 (36.154)
  Percentage of time below target range | 20.76 (36.587) | 18.34 (35.778) | 25.44 (40.120) | 29.39 (42.670) | 32.76 (43.780) | 17.89 (36.836)

4. Secondary Outcome: Number of Participants With Hgb in the Target Range at Week 24
Description: The number of participants with Hgb in the target range of 10.0 to 11.5 g/dL at Week 24 was recorded for each arm.
Time Frame: Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 24 | 18 | 27 | 26 | 24 | 11
Participants | 14 | 13 | 16 | 10 | 15 | 8

5. Secondary Outcome: Number of Participants Reaching Pre-defined Hgb Stopping Criteria
Description: The number of participants who reached the Hgb stopping criteria of Hgb concentration <7.5 g/dL were presented.
Time Frame: Up to 24 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 39 | 38 | 39 | 38 | 39 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Observed Change From Baseline in Erythropoietin (EPO)
Description: Blood samples for control arm were collected on Day 1 (pre-dose), Week 4 (5-15 minutes post-dose), Week 8 (pre-dose), Week 12 (pre-dose), Week 16 (pre-dose), Week 20 (pre-dose, 5-15 minutes post-dose), Week 24 (pre-dose), and Week 28 (pre-dose) for EPO measurement. Blood samples for GSK1278863 arms were collected on Day 1 (pre-dose), Week 4 (6-12 hours post-dose), Week 4 (7-13, 8-14, 9-15, hours post-dose), Week 8 (pre-dose), Week 12 (pre-dose), Week 16 (pre-dose), Week 20 (pre-dose, 3 hour post-dose) Week 24 (pre-dose), and Week 28 (pre-dose) for EPO measurement. The maximum observed change from baseline in EPO was recorded for each arm. Baseline value for EPO is the pre-dose value on Day 1. Change from Baseline in EPO was calculated as the individual post-dose values minus the Baseline value.
Time Frame: Baseline (Day 1) to Week 28
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: international units(IU)/Liter (L)
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 36 | 37 | 37 | 37 | 36 | 16
international units(IU)/Liter (L) | 1946.45 (8456.313) | 48.86 (117.050) | 36.63 (35.485) | 84.53 (225.768) | 82.00 (99.660) | 24.63 (235.820)

7. Secondary Outcome: Maximum Observed Percent Change From Baseline in Vascular Endothelial Growth Factor (VEGF)
Description: Blood samples for control arm were collected on Day 1 (pre-dose), Week 4 (5-15 minutes post-dose), Week 8 (pre-dose), Week 12 (pre-dose), Week 16 (pre-dose), Week 20 (pre-dose, 5-15 minutes post-dose), Week 24 (pre-dose), and Week 28 (pre-dose) for VEGF measurement. Blood samples for GSK1278863 arms were collected on Day 1 (pre-dose), Week 4 (6-12 hours post-dose), Week 4 (7-13, 8-14, 9-15, hours post-dose), Week 8 (pre-dose), Week 12 (pre-dose), Week 16 (pre-dose), Week 20 (pre-dose, 3 hour post-dose) Week 24 (pre-dose), and Week 28 (pre-dose) for VEGF measurement. The maximum observed percent change from Baseline in VEGF was recorded for each arm. Baseline value for VEGF is the pre-dose value on Day 1. Percent change from Baseline was calculated as 100 multiplied by exponential of mean change in log scale minus 1.
Time Frame: Baseline (Day 1) to Week 28
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 36 | 37 | 37 | 37 | 36 | 16
Percent change | 36.02 [16.45 to 58.87] | 36.92 [19.33 to 57.11] | 41.73 [22.65 to 63.77] | 54.91 [37.38 to 74.69] | 50.65 [31.88 to 72.10] | 50.97 [21.49 to 87.60]

8. Secondary Outcome: Population Plasma PK Parameters of GSK1278863 and Metabolites
Description: Blood samples were collected for individual plasma GSK1278863and metabolite (GSK2391220, GSK2499166, GSK2531403, GSK2531400, GSK2531399, and GSK2531398) concentrations measurement on Day (D) 1 (pre-dose [PrD), at Week (W) 4 (6-12, 7-13, 8-14, and 9-15 hour [hr] post-dose [PoD), and at W20 (PrD, 1, 2, and 3 hour PoD). Pharmacokinetic population: All participants from whom a PK sample has been obtained and analyzed.
Time Frame: Day 1, Week 4, and Week 20
Population: Pharmacokinetic Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points; thus, the overall number of participants analyzed reflects everyone in the pharmacokinetic population
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 19
nanograms (ng)/milliliter (mL)
  GSK1278863, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK1278863, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 6.3 (10.04) | 9.3 (19.06) | 7.7 (18.46) | 25.4 (53.37) | 9.0 (18.80)
  GSK1278863, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 10.6 (25.15) | 16.3 (57.24) | 8.7 (19.85) | 19.9 (42.65) | 8.0 (16.92)
  GSK1278863, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 7.5 (16.80) | 8.1 (23.76) | 5.6 (11.75) | 12.7 (28.60) | 4.6 (6.87)
  GSK1278863, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 6.8 (14.53) | 4.6 (10.49) | 4.4 (9.19) | 11.3 (25.36) | 11.2 (33.59)
  GSK1278863, W20, PrD, n=23, 28, 27, 23, 14 | 2.3 (6.44) | 0.7 (2.55) | 0.9 (2.82) | 7.9 (30.99) | 6.6 (20.22)
  GSK1278863, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 25.9 (35.74) | 37.6 (53.77) | 88.2 (153.06) | 58.5 (85.91) | 65.2 (127.21)
  GSK1278863, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 34.2 (31.76) | 52.4 (53.32) | 62.8 (85.37) | 82.7 (117.97) | 63.3 (102.15)
  GSK1278863, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 43.6 (58.36) | 39.2 (44.59) | 44.1 (70.53) | 71.2 (110.91) | 65.8 (100.80)
  GSK2391220, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK2391220, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 9.1 (6.68) | 12.9 (8.32) | 18.5 (13.72) | 20.1 (12.32) | 21.3 (17.34)
  GSK2391220, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 5.1 (4.22) | 6.7 (5.51) | 10.3 (8.55) | 10.9 (6.37) | 13.1 (12.44)
  GSK2391220, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 3.8 (3.66) | 4.5 (4.16) | 7.4 (6.44) | 7.4 (4.51) | 7.2 (6.97)
  GSK2391220, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 3.3 (3.76) | 3.3 (3.15) | 5.3 (4.86) | 5.4 (3.63) | 6.6 (5.72)
  GSK2391220, W20, PrD, n=23, 28, 27, 23, 14 | 5.0 (7.72) | 3.2 (4.97) | 4.1 (5.84) | 4.6 (9.29) | 3.5 (6.69)
  GSK2391220, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 3.9 (5.59) | 2.7 (3.60) | 4.3 (4.90) | 5.0 (8.10) | 2.6 (3.64)
  GSK2391220, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 5.4 (5.58) | 4.5 (4.96) | 6.5 (6.93) | 8.1 (10.33) | 4.9 (4.08)
  GSK2391220, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 5.3 (4.64) | 5.0 (5.26) | 7.3 (6.69) | 8.2 (6.52) | 6.1 (4.92)
  GSK2487818, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK2487818, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 3.1 (2.82) | 4.1 (4.47) | 5.7 (6.31) | 7.2 (6.57) | 5.2 (4.66)
  GSK2487818, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 1.8 (1.75) | 2.6 (3.81) | 3.5 (4.55) | 4.1 (3.73) | 3.7 (4.61)
  GSK2487818, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 1.5 (1.67) | 1.9 (3.21) | 2.7 (3.58) | 2.7 (2.44) | 1.7 (1.68)
  GSK2487818, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 1.4 (1.88) | 1.5 (2.46) | 1.9 (2.85) | 1.9 (1.92) | 1.9 (2.21)
  GSK2487818, W20, PrD, n=23, 28, 27, 23, 14 | 1.2 (3.38) | 0.5 (1.05) | 0.7 (1.28) | 1.3 (4.09) | 0.7 (1.84)
  GSK2487818, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 2.0 (3.82) | 1.3 (1.73) | 2.7 (3.97) | 3.4 (5.88) | 1.0 (1.34)
  GSK2487818, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 3.8 (4.58) | 3.6 (4.36) | 5.0 (5.82) | 6.3 (8.04) | 3.7 (3.28)
  GSK2487818, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 3.9 (3.49) | 4.3 (4.76) | 5.7 (5.28) | 6.5 (5.05) | 5.0 (4.43)
  GSK2506102, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK2506102, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 3.2 (1.98) | 4.9 (2.68) | 6.6 (4.16) | 7.6 (4.30) | 9.0 (6.19)
  GSK2506102, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 1.8 (1.31) | 2.5 (1.71) | 3.7 (2.60) | 4.1 (2.15) | 5.4 (4.10)
  GSK2506102, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 1.3 (1.07) | 1.6 (1.16) | 2.6 (1.94) | 2.9 (1.68) | 2.9 (2.24)
  GSK2506102, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 1.1 (1.16) | 1.2 (0.88) | 1.9 (1.52) | 2.1 (1.23) | 2.7 (2.04)
  GSK2506102, W20, PrD, n=23, 28, 27, 23, 14 | 2.3 (1.99) | 1.9 (2.05) | 2.3 (2.09) | 2.6 (2.87) | 2.2 (2.87)
  GSK2506102, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 1.4 (1.27) | 1.1 (1.40) | 1.4 (1.22) | 1.8 (2.12) | 1.4 (1.57)
  GSK2506102, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 1.5 (1.25) | 1.2 (1.24) | 1.8 (1.72) | 2.2 (2.53) | 1.6 (1.37)
  GSK2506102, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 1.4 (1.12) | 1.3 (1.26) | 1.9 (1.53) | 2.1 (1.66) | 1.7 (1.42)
  GSK2531398, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK2531398, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 3.4 (2.46) | 4.9 (3.11) | 6.9 (4.52) | 8.0 (4.87) | 7.9 (5.75)
  GSK2531398, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 2.0 (1.72) | 2.7 (2.41) | 4.0 (2.97) | 4.5 (2.70) | 4.9 (4.05)
  GSK2531398, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 1.5 (1.46) | 1.8 (1.86) | 2.9 (2.30) | 3.1 (1.95) | 2.5 (1.78)
  GSK2531398, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 1.4 (1.58) | 1.4 (1.49) | 2.1 (1.99) | 2.2 (1.38) | 2.3 (1.42)
  GSK2531398, W20, PrD, n=23, 28, 27, 23, 14 | 1.5 (2.31) | 1.2 (2.03) | 1.4 (1.93) | 1.6 (3.80) | 1.2 (2.67)
  GSK2531398, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 1.3 (1.89) | 1.0 (1.34) | 1.6 (1.81) | 2.0 (3.58) | 1.0 (1.45)
  GSK2531398, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 2.1 (2.24) | 1.9 (2.09) | 2.9 (3.28) | 3.5 (4.69) | 2.1 (1.79)
  GSK2531398, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 2.3 (2.04) | 2.2 (2.22) | 3.3 (2.89) | 3.8 (3.10) | 2.8 (2.34)
  GSK2531401, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.02)
  GSK2531401, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 9.9 (8.00) | 14.7 (10.02) | 22.2 (14.71) | 24.5 (18.27) | 29.1 (24.55)
  GSK2531401, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 5.4 (4.49) | 7.1 (5.53) | 11.8 (8.49) | 13.1 (9.50) | 17.3 (16.03)
  GSK2531401, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 4.0 (3.63) | 4.5 (3.50) | 8.1 (5.74) | 9.0 (7.05) | 10.1 (10.61)
  GSK2531401, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 3.3 (3.36) | 3.2 (2.35) | 5.9 (4.66) | 6.3 (4.90) | 8.7 (8.72)
  GSK2531401, W20, PrD, n=23, 28, 27, 23, 14 | 7.7 (7.71) | 7.3 (7.34) | 7.9 (7.37) | 9.3 (10.95) | 7.2 (10.04)
  GSK2531401, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 4.2 (4.52) | 4.0 (6.77) | 4.7 (4.18) | 5.6 (7.48) | 4.5 (5.44)
  GSK2531401, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 4.2 (4.44) | 3.6 (4.50) | 4.8 (4.08) | 6.1 (8.21) | 4.4 (4.41)
  GSK2531401, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 4.1 (4.07) | 3.6 (4.55) | 5.0 (4.64) | 5.5 (5.38) | 4.5 (4.28)
  GSK2531403, D1, PrD, n=39, 40, 39, 40, 18 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  GSK2531403, W4, 6-12 hr PoD, n=36, 37, 37, 35, 15 | 11.4 (7.47) | 17.0 (9.89) | 23.1 (15.22) | 25.4 (14.25) | 28.8 (21.46)
  GSK2531403, W4, 7-13 hr PoD, n=36, 37, 35, 35, 15 | 6.3 (4.84) | 8.6 (6.43) | 13.1 (9.73) | 13.9 (7.66) | 17.4 (14.72)
  GSK2531403, W4, 8-14 hr PoD, n=35, 37, 36, 35, 15 | 4.7 (4.23) | 5.7 (4.63) | 9.3 (7.37) | 9.6 (5.50) | 9.9 (9.05)
  GSK2531403, W4, 9-15 hr PoD, n=35, 36, 36, 35, 15 | 4.1 (4.60) | 4.1 (3.41) | 6.7 (5.50) | 6.9 (4.25) | 8.9 (7.79)
  GSK2531403, W20, PrD, n=23, 28, 27, 23, 14 | 7.8 (8.53) | 6.0 (8.08) | 6.7 (6.74) | 7.8 (11.14) | 6.2 (8.78)
  GSK2531403, W20, 1 hr PoD, n=23, 27, 27, 24, 13 | 4.9 (5.56) | 3.8 (4.88) | 5.0 (4.71) | 6.2 (8.65) | 4.0 (4.80)
  GSK2531403, W20, 2 hr PoD, n=23, 27, 27, 24, 13 | 5.7 (5.43) | 4.7 (4.91) | 6.8 (6.54) | 8.5 (10.83) | 5.5 (4.58)
  GSK2531403, W20, 3 hr PoD, n=23, 27, 27, 24, 14 | 5.5 (4.52) | 5.1 (5.18) | 7.4 (6.43) | 8.4 (6.86) | 6.5 (5.14)

9. Secondary Outcome: Percent Change From Baseline in Hepcidin at Week 24
Description: Hepcidin is a regulator of iron metabolism. Baseline value for transferrin saturation is the pre-dose value on Day 1. Percent change from Baseline was calculated as 100 multiplied by exponential of mean change in log scale minus 1.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 32 | 20 | 29 | 26 | 25 | 14
Percent change | 3.63 [-20.39 to 34.89] | -17.39 [-42.36 to 18.40] | -11.85 [-26.47 to 5.67] | -30.28 [-48.08 to -6.37] | -6.91 [-28.69 to 21.52] | -42.13 [-62.82 to -9.95]

10. Secondary Outcome: Change From Baseline in Ferritin at Week 24
Description: Baseline value for ferritin is the pre-dose value on Day 1. Change from Baseline in ferritin was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Micrograms/Liter
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 33 | 20 | 29 | 27 | 25 | 14
Micrograms/Liter | 56.8 (214.27) | -29.4 (357.10) | -50.4 (408.99) | -95.6 (304.61) | -20.2 (227.34) | -125.2 (354.64)

11. Secondary Outcome: Change From Baseline in Transferrin at Week 24
Description: Baseline value for transferrin is the pre-dose value on Day 1. Change from Baseline in transferrin was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: grams (g)/Liter (L)
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 33 | 20 | 29 | 27 | 25 | 14
grams (g)/Liter (L) | -0.133 (0.2903) | 0.238 (0.3709) | 0.198 (0.2891) | 0.226 (0.2706) | 0.249 (0.3213) | 0.393 (0.3165)

12. Secondary Outcome: Percent Change From Baseline in Transferrin Saturation at Week 24
Description: Transferrin saturation is measured as a percentage, it is the ratio of serum iron and total iron-binding capacity, multiplied by 100. Baseline value for transferrin saturation is the pre-dose value on Day 1. Percent change from Baseline =: 100*(exp(Mean change log scale)-1).
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 32 | 20 | 29 | 27 | 25 | 14
Percent change | -9.0 [-27.3 to 13.9] | -3.7 [-22.9 to 20.4] | -12.1 [-23.4 to 0.9] | -8.3 [-22.9 to 9.0] | 8.2 [-7.7 to 26.8] | -2.5 [-16.0 to 13.2]

13. Secondary Outcome: Change From Baseline in Total Iron at Week 24
Description: Baseline value for total iron is the pre-dose value on Day 1. Change from Baseline in total iron was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles/Liter
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 33 | 20 | 29 | 27 | 25 | 14
Micromoles/Liter | -0.8 (7.64) | 0.9 (9.75) | 0.3 (5.20) | 0.2 (6.51) | 2.0 (3.96) | 1.6 (3.18)

14. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity at Week 24
Description: Total iron-binding capacity is a medical laboratory test that measures the blood's capacity to bind iron with transferrin. Baseline value for total iron binding capacity is the pre-dose value on Day 1. Change from Baseline in total iron binding capacity was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles/Liter
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 32 | 20 | 29 | 27 | 25 | 14
Micromoles/Liter | -2.0 (4.48) | 6.0 (7.93) | 4.2 (6.79) | 6.6 (5.75) | 4.8 (6.25) | 6.2 (6.44)

15. Secondary Outcome: Change From Baseline in Reticulocyte Hemoglobin at Week 24
Description: Baseline value for reticulocyte hemoglobin is the pre-dose value on Day 1. Change from Baseline in reticulocyte hemoglobin was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 30 | 20 | 29 | 26 | 24 | 12
Picogram | -0.19 (1.610) | -0.28 (1.948) | -0.62 (2.046) | -0.42 (1.458) | -0.51 (1.377) | -0.63 (1.119)

16. Secondary Outcome: Change From Baseline in Hematocrit at Week 24
Description: Hematocrit is the ratio of the volume of red blood cells to the total volume of blood. Baseline value for hematocrit is the pre-dose value on Day 1. Change from Baseline in hematocrit was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 30 | 20 | 29 | 28 | 26 | 13
Ratio | -0.0028 (0.04358) | -0.0096 (0.04073) | 0.0020 (0.03579) | 0.0043 (0.04254) | -0.0021 (0.02678) | 0.0108 (0.03557)

17. Secondary Outcome: Change From Baseline in Red Blood Cells at Week 24
Description: Baseline value for red blood cells is the pre-dose value on Day 1. Change from Baseline in red blood cells was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/Liter
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 30 | 20 | 29 | 28 | 26 | 13
10^12 cells/Liter | 0.01 (0.460) | -0.06 (0.396) | 0.04 (0.374) | 0.07 (0.399) | 0.03 (0.300) | 0.17 (0.366)

18. Secondary Outcome: Change From Baseline in Reticulocyte Count at Week 24
Description: A reticulocyte count is a blood test that measures the percentage of reticulocytes in the blood. Reticulocytes are slightly immature red blood cells. Baseline value for reticulocyte count is the pre-dose value on Day 1. Change from Baseline in reticulocyte count was calculated as the Week 24 value minus the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: ITT Population. Only participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in blood
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Number analyzed (Participants) | 31 | 20 | 30 | 28 | 26 | 12
Percentage of reticulocytes in blood | 0.40 (0.663) | 0.16 (1.162) | 0.18 (0.571) | 0.03 (0.684) | -0.15 (0.838) | 0.10 (0.527)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until the follow up contact (up to 28 weeks).
Description: Post baseline SAEs and non-serious AEs were reported for the Safety population which consisted of all participants who received at least one dose of study drug.
Arm/Group | Control | GSK1278863 4 mg | GSK1278863 6 mg | GSK1278863 8 mg | GSK1278863 10 mg | GSK1278863 12 mg
Serious Adverse Events (participants affected / at risk) | 11/39 | 10/39 | 8/40 | 8/39 | 11/40 | 1/19
Other Adverse Events (participants affected / at risk) | 17/39 | 28/39 | 17/40 | 25/39 | 21/40 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=39) | GSK1278863 4 mg (N=39) | GSK1278863 6 mg (N=40) | GSK1278863 8 mg (N=39) | GSK1278863 10 mg (N=40) | GSK1278863 12 mg (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dialysis related complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Steal syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=39) | GSK1278863 4 mg (N=39) | GSK1278863 6 mg (N=40) | GSK1278863 8 mg (N=39) | GSK1278863 10 mg (N=40) | GSK1278863 12 mg (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 2 | 1 | 1 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Retinal artery embolism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 2 | 7 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 3 | 2 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 2 | 0
Asthenia (General disorders) | 0 | 2 | 3 | 0 | 0 | 0 — General disorders and administration site conditions
Chills (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 — General disorders and administration site conditions
Face oedema (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 — General disorders and administration site conditions
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 — General disorders and administration site conditions
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 1 | 0 | 2 | 2 | 1 | 0 — General disorders and administration site conditions
Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 — General disorders and administration site conditions
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 5 | 6 | 3 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 0
Dialysis related complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 1 | 3 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 0 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 4 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 1 | 6 | 0 | 2 | 4 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.